CLINICAL TRIAL: NCT05674409
Title: Evaluating the Efficacy of Telehealth-Delivered Brief Family Involved Treatment (B-FIT) for Alcohol Use Disorder Among Veterans
Brief Title: Brief Family Involved Treatment Telehealth
Acronym: B-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Julianne Flanagan, Associate Professor, Licensed Clinical Psychologist, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00121552; R01AA029679 (NIH)
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Behavioral Therapy; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy + Brief Family-Involved Treatment (Experimental): Approximately half of enrolled veterans and their treatment companion will be randomly assigned to the experimental group. The identified veteran participant wil receive 12 sessions of Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD). In addition, both the identified veteran and their treatment companion will receive an additional 3 sessions of Brief Family-Involved Treatment (B-FIT).
  B-FIT is a manualized, 3-session AUD intervention, designed to be implemented in combination with any existing alcohol treatment program.
  Interventions: Behavioral: Brief Family-Involved Treatment (B-FIT); Behavioral: Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD)
- Cognitive Behavioral Therapy (Active Comparator): Approximately half of enrolled veterans and their treatment companion will be randomly assigned to the active comparator group. The identified veteran participant wil receive 12 sessions of Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD).
  Interventions: Behavioral: Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD)

INTERVENTIONS:
Behavioral: Brief Family-Involved Treatment (B-FIT) — Brief Family-Involved Treatment (B-FIT) is a manualized, 3-session intervention for Alcohol Use Disorder (AUD). Designed to be implemented in combination with any existing alcohol treatment program, the goals of B-FIT are to (1) increase reinforcement for AUD treatment engagement, (2) increase positive rewards from drinking reductions, and (3) decrease drinking cues by decreasing negative communication and increasing positive communication.
  Arms: Cognitive Behavioral Therapy + Brief Family-Involved Treatment
Behavioral: Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD) — Participants will receive 12 sessions of Cognitive Behavioral Therapy for Alcohol Use Disorder (CBT for AUD).

SUMMARY:
Improving alcohol use disorder (AUD) treatment among Veterans is a national public health problem. The rate of AUD among Veterans is twice that of civilians, with up to 50% of Veterans having AUD. Family-based AUD programs are rarely undertaken in busy treatment clinics, and Veterans with problem drinking behavior or AUD are commonly excluded from couple therapies. As a result, there is a need to develop effective family AUD treatments that are both brief and highly accessible to Veterans.

The purpose of this study is to evaluate a new treatment add-on called Brief Family-Involved Treatment (B-FIT), which will be delivered via telehealth among Veterans engaged in alcohol-based treatment/therapy.

This study is an 12-week, Stage-II, open randomized controlled trial examining B-FIT in combination with treatment as usual (TAU), (in this case B-FIT+ Cognitive Behavioral Therapy treatment) as compared to TAU alone (CBT treatment).Veterans and their treatment companion (family member, partner, friend) will complete weekly assessments during the treatment phase in addition to 3 & 6 month follow-up assessments, all via telehealth.

DETAILED DESCRIPTION:
Improving alcohol use disorder (AUD) treatment among Veterans is a national public health priority. The prevalence of AUD among Veterans is twice that of civilians, with up to 50% of Veterans meeting diagnostic criteria for lifetime AUD. Although one in 6 Veterans has an AUD diagnosis in their medical record, substantial barriers to accessing evidence-based AUD treatment persists in this population. While adaptive family support is a critical ingredient to effective AUD treatment and drinking reductions, maladaptive family functioning interferes with AUD recovery and is a precipitant of relapse. Family participation in AUD treatment has the ability to optimize engagement and outcomes.

Family-based AUD programs are rarely undertaken in busy treatment clinics, and Veterans with problem drinking behavior or AUD are commonly excluded from couple therapies. There is an urgent need to develop efficacious family AUD treatments that are both brief and highly accessible to Veterans. Brief Family-Involved Treatment (B-FIT) delivered via telehealth is an intervention distilled from the robustly evidence-based Alcohol Behavioral Couple Therapy (ABCT) model. Designed to be implemented in combination with any existing alcohol treatment program, the goals of B-FIT are to (1) increase reinforcement for AUD treatment engagement, (2) increase positive rewards from drinking reductions, and (3) decrease drinking cues by decreasing negative communication and increasing positive communication.

The objective of the proposed Stage II study is to evaluate the efficacy of B-FIT delivered via telehealth among Veterans enrolled manualized treatment for AUD (Cognitive Behavioral Therapy, CBT). We will also examine putative individual and family characteristics that mediate treatment outcomes. To accomplish this, we will employ an open randomized controlled design and examine standardized, repeated, dependent measures of change. Veterans and a family member (or concerned partner/friend) will be randomly assigned (matched on age, sex and baseline alcohol consumption) to receive B-FIT in combination with TAU (CBT) or TAU alone. A total of 200 veterans and their treatment companions will be enrolled in this study (N=400).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 200 Veterans and a family member, plus their treatment companion, a concerned partner or friend (total N=400; 50% women veterans) aged 21 or older.

Inclusion criteria for Veterans require that they:

1. Meet diagnostic criteria for current moderate to severe alcohol use disorder (AUD) with 2 or more heavy drinking days (>5 for men, >4 for women) in the 60 days prior to enrollment
2. Have an adult family member/treatment companion who is willing to participate
3. Demonstrate cognitive functioning sufficient to provide informed consent and participate accurately (≥ 26 on the Mini-Mental Status Exam [MMSE])
4. Maintain a stable dose of psychotropic medications for at least 4 weeks before enrollment. Concurrent drug use disorders are acceptable provided alcohol is the Veteran's primary substance of choice. Drug use will be measured weekly and controlled for in statistical analyses if needed.

Inclusion criteria for the family member/treatment companion require that they:

1. Are not receiving or seeking treatment for their own alcohol or drug problem
2. Report total Alcohol Use Disorders Identification Test (AUDIT) scores <8
3. Report total Drug Abuse Screening Test (DAST-10) scores <3.

Exclusion Criteria:

Exclusion criteria for all participants include:

1. History of or current psychotic or bipolar disorder
2. Alcohol withdrawal (Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) score >8)
3. Current suicidal or homicidal ideation and intent
4. Severe or unilateral violence in the past 6 months as measured by the Revised Conflict Tactics Scale (CTS2) (consistent with extant dyadic treatment literature).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Family functioning | From baseline to week 12
  Change in family functioning as measured by the Brief Family Assessment Measure-III (Brief FAM-III)
Change in Alcohol Consumption | From baseline to week 12
  Change in percent days abstinent, as measured by the Alcohol Timeline Followback (TLFB)
Change in percent days drinking | From baseline to week 12
  Change in percent days drinking, as measured by the Alcohol Timeline Followback (TLFB)
Change in drinks per drinking day | From baseline to week 12
  Change in drinks per drinking day , as measured by the Alcohol Timeline Followback (TLFB)
Alcohol problem severity | From baseline to week 12
  Change in Alcohol problem severity as measured by the Alcohol Use Disorders Identification Test (AUDIT)
Change in alcohol craving | From baseline to week 12
  Change in alcohol craving as measured by the Penn Alcohol Craving Scale (PACS)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States